CLINICAL TRIAL: NCT07114575
Title: Spatiotemporal Characteristics of Gait at Different Walking Speeds in Individuals With Stroke
Brief Title: Gait Characteristics at Different Speeds in Individuals With Stroke
Status: Recruiting | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Murat Akıncı, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: VR01
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: stroke; spatial; temporal; walking; analysis
MeSH Terms: conditions — Stroke | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Self Selected Speed: Participants in this group will perform the gait analysis at their preferred comfortable walking speed.
  Interventions: Other: Gait Analysis
- Slow Walking Speed: Participants in this group will walk at a speed approximately 25% slower than their comfortable walking speed.
  Interventions: Other: Gait Analysis
- Fast Walking Speed: Participants in this group will walk at a speed approximately 25% faster than their comfortable walking speed.
  Interventions: Other: Gait Analysis

INTERVENTIONS:
Other: Gait Analysis — All participants will undergo gait analysis at three different walking speeds.

SUMMARY:
Stroke is the second leading cause of death and the third leading cause of death combined with disability worldwide. Despite improved recognition and management of stroke risk factors, the risk of stroke has increased by 50% in the last two decades due to increased life expectancy, currently affecting one in every four individuals. If this trend continues, by 2030, it is estimated that 12 million people will die from stroke, and 70 million will live with its consequences.

Stroke leads to significant changes in the spatiotemporal parameters of gait. Spatial parameters include step length, stride length, and step width, while temporal parameters comprise cadence, stance phase, double support phase (DSP), and swing phase. Gait speed, incorporating both spatial and temporal elements, is classified as a spatiotemporal parameter. Compared to healthy individuals, people post-stroke tend to have increased DSP and stance phases, shortened step lengths, and widened step widths. Asymmetries between the paretic and non-paretic limbs further disrupt gait symmetry.

Previous studies have shown that during prolonged walking tasks such as the 6-minute walk test, both gait speed and symmetry deteriorate in the later stages, potentially due to fatigue. However, changes in walking speed itself may also influence gait symmetry. From this perspective, the aim of this study is to investigate how spatiotemporal gait parameters vary across different walking speeds in individuals with stroke.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death and disability worldwide, with increasing prevalence due to longer life expectancy, despite improved recognition and management of risk factors. Stroke-related impairments, particularly in gait, significantly affect individuals' independence and quality of life. Post-stroke gait is commonly characterized by altered spatiotemporal parameters, including reduced step length, increased double support phase, asymmetry between paretic and non-paretic limbs, and reduced walking speed.

This descriptive study aims to investigate how different walking speeds affect the spatiotemporal gait parameters in individuals with stroke. Specifically, the study will examine walking at comfortable, slow (-25%), and fast (+25%) speeds using an instrumented treadmill (C-Mill). The target population includes adult individuals (18+) diagnosed with hemiplegia (ICD-10: G81), who are able to ambulate with or without assistance (Functional Ambulation Classification ≥2).

Spatiotemporal gait parameters, including step length, step width, cadence, stance and swing phases, and double support time, will be collected for both paretic and non-paretic limbs. These parameters will be assessed at three different walking speeds. In addition to gait analysis, functional status will be evaluated using the Functional Ambulation Classification (FAC), Berg Balance Scale (BBS), and the lower extremity section of the Fugl-Meyer Assessment (FMA-LE). Demographic and clinical information will also be recorded.

Participants will first walk at their comfortable speed to familiarize themselves with the treadmill and to determine baseline parameters. After a 2-minute warm-up walk, a 2-minute data collection phase will follow. The same procedure will be repeated at the slow and fast walking speeds. Gait symmetry and changes in temporal-spatial parameters across walking speeds will be analyzed to explore the influence of speed variation, particularly regarding the mechanisms underlying gait asymmetry and fatigue.

This research will provide insight into how walking speed modulates gait parameters in stroke survivors and may contribute to developing more targeted gait training strategies in neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Having an ICD-10 diagnosis code of G.81 Hemiplegia
* Ability to walk with or without assistance (Functional Ambulation Classification score of 2 or higher)

Exclusion Criteria:

* Presence of any known additional neurological or orthopedic condition that may affect walking
* Inability to complete the tests due to cognitive and/or physical reasons
* Inability to complete the analysis at walking speeds increased or decreased by 25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Stance Phase | Baseline
  Stance phase of hemiplegic side during walking. This outcome will be obtained as a result of the gait analysis
Hemiplegic Side Step Length | Baseline
  Step legth of hemiplegic side during walking. This outcome will be obtained as a result of the gait analysis
Double Support Phase | Baseline
  Double support phase during walking. This outcome will be obtained as a result of the gait analysis

SECONDARY OUTCOMES:
Stride Length | Baseline
  Stride length during walking. This outcome will be obtained as a result of the gait analysis.

OTHER OUTCOMES:
Fugl Meyer Lower Extremity | Baseline
  This is a widely used, reliable, and valid test to evaluate motor impairments of the paretic upper and lower extremities in stroke patients. Each item on the scale is scored as 0: unable to perform, 1: partially successful performance, and 2: fully successful performance. Higher scores indicate better motor function. In our study, the 34-point lower extremity section will be used.
Berg Balance Scale | Baseline
  The scale consists of 14 items and assesses the patient's ability to maintain balance (during static or various functional movements) over a certain period. Each item is scored from 0 to 4: 0 points indicate inability to complete the task, while 4 points indicate independent completion of the task. The total maximum score is 56. Scores between 0-20 indicate balance impairment, 21-40 indicate acceptable balance, and 41-56 indicate good balance.
Functional Ambulation Category | Baseline
  The scale, which is valid and reliable for patients who develop hemiparesis after stroke, classifies walking ability into six levels based on the amount of physical assistance required (8). A score of 0 indicates that the patient needs assistance from two people to walk, while a score of 5 indicates independent walking in all environments, including stairs.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, None Selected, Turkey (Türkiye)